CLINICAL TRIAL: NCT03783234
Title: 3-level Triage Assessment and National Early Warning Score as Predictor for Mortality, Hospital Admission and ED Readmission for Older Frailty Patients in the ED
Brief Title: Triage Assessment and NEWS-score as Risk Predictor in Older Frailty Adults in the ED
Status: Completed | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: City of Espoo (Unknown); University of Helsinki (Other)
Responsible Party: Principal Investigator, Janne Alakare, Senior physician in Emergency Medicine, Helsinki University Central Hospital
Other Study IDs: HUS/278/2018
Record Dates: First submitted 2018-12-19; First posted 2018-12-20 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Frailty; Aged; Triage
Keywords: Emergency triage
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Older Adult Patients: ED patients age of ≥ 75 who have nurse assessed Clinical Frailty Scale ≥ 4.

SUMMARY:
Emergency Department Triage Systems have not been shown to sufficiently recognize frail elderly patients in need of urgent assessment and care. In this prospective, observational study the performance of the 3-level triage system and the National Early Warning Score (NEWS) 2 are assessed (separately and combined) for predicting adverse outcomes in older frailty patients visiting in the ED. Observational data for this study is gathered as part of GAOPS - main study (ClinicalTrials.gov Identifier: NCT03751319).

ELIGIBILITY:
Inclusion Criteria:

* "Clinical Frailty Scale" minimum 4 estimated at the arrival to the ED by nurse

Exclusion Criteria:

• Non-resident of the counties (City of Espoo, Kirkkonummi, Kauniainen) of the hospital district.

Min Age: 75 Years | Sex: All
Age Groups: Older Adult
Study Population: Residents of aforementioned counties, aged over 75 years, who attend the Emergency department and have clinical frailty scale minimum 4.
Sampling Method: Non-Probability Sample
Enrollment: 1711 (Actual)
Dates: Start 2018-12-11 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2020-10-28 (Actual)

PRIMARY OUTCOMES:
Mortality | 30 days
  Mortality during the 30 day follow-up

SECONDARY OUTCOMES:
Hospital admission | Day 0
  Admission to hospital from the Emergency Department
ICU/HDU admission | Day 0
  Admission to the Intensive Care Unit or High Dependency Unit from the Emergency Department
Readmission in the ED | Hour 72, Day 30
  Re-visits to the ED after the index-visit

CONTACTS AND LOCATIONS:
Overall Officials: Veli-Pekka Harjola, Study Director — Department of Emergency Medicine and Services, Helsinki University Hospital; Janne Alakare, MD, Principal Investigator — Department of Emergency Medicine and Services, Helsinki University Hospital
Locations (1):
- Helsinki University Central Hospital, Jorvi, Espoo, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kemp K, Alakare J, Harjola VP, Strandberg T, Tolonen J, Lehtonen L, Castren M. National Early Warning Score 2 (NEWS2) and 3-level triage scale as risk predictors in frail older adults in the emergency department. BMC Emerg Med. 2020 Oct 28;20(1):83. doi: 10.1186/s12873-020-00379-y. PMID 33115446
- See also: Full text — https://bmcemergmed.biomedcentral.com/articles/10.1186/s12873-020-00379-y